CLINICAL TRIAL: NCT06051916
Title: Post-operative Residual Voiding Volume Following Bulking and Vaginal Prolapse Surgery and Impact on In-hospital Stay
Acronym: POUR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Martin Rudnicki, Professor, Odense University Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Odense University Hospital SDU
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Surgery-Complications
Keywords: surgery; complication

STUDY DESIGN:
Intervention Model Description: Group A receives a strict voiding trial and group B receives a minimalistic voiding trial. In both groups the patient's catheter is removed at the operation room before returning to the gynecological ward.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group B (Active Comparator): Group B is the intervention group with minimalistic voiding trial. The patients in this group need to have one spontaneous voiding before discharge with the sensation of normal voiding, meaning there is no measurement of the voiding volume or residual volume.
  Interventions: Other: residual urine
- Group A (No Intervention): Group A is the control group and presents the current procedures with strict voiding trial. The bladder is scanned before voiding to determine the bladder volume, and the voiding volume is measured. If the voiding volume is >150 ml and the residual volume is <200 ml, the patient can be discharged. If no acceptable residual volume is reached, the patient will be instructed in intermittent catheterization

INTERVENTIONS:
Other: residual urine — The study includes two group, A and B. Se previously
  Arms: group B

SUMMARY:
Post operative urinary retention is a commonly observed complication following women undergoing urogynecology surgery.

The trial includes patients undergoing bulking and vaginal prolapse surgery, who are randomized in two postoperative groups prior to surgery in order to test two void regimes. One group includes a strict voiding regime, where patients are discharged when voiding volume is minimum 150 ml and residual volume is maximum 200 ml. Comparatively, the minimalistic voiding group discharge patients after one spontaneous voiding, independent of voiding volume and residual volume.

The primary aim of this study is to evaluate time to discharge in two different voiding trials techniques (strict vs minimalistic) after anterior, posterior or vaginal vault prolapse surgery as well as bulking surgery. Secondly, to register the development of postoperative urinary tract infection, urine retention, gynecological pain and patients' calls to the gynecological ward after discharge.

DETAILED DESCRIPTION:
Project description Aim The primary aim of this study is to evaluate time to discharge in two different voiding trials techniques (strict vs minimalistic) after anterior, posterior or vaginal vault prolapse surgery as well as bulking surgery.

Secondly, to evaluate the frequency of postoperative urinary tract infection, urine retention and pain as well as patients' calls to the gynecological ward after discharge.

Hypothesis The hypothesis is that the intervention group (minimalistic trial) will have an earlier discharge and fewer complications compared to the other group (strict trial).

Materials and methods The study will be performed as a two-armed parallel randomized controlled trial. Relevant patients at Odense University Hospital will be informed about the study at the preoperative consultation.

Prior to inclusion all patients are provided with verbal and written information regarding the study protocol and they give their informed consent. All patients will be randomized by a computer-generated list in a ratio of 1:1 to either strict or minimalistic regime. Randomization is done using Redcap. An independent statistician generates the random allocation sequence. The study will be blinded for the operating doctor.

Group A receives a strict voiding trial and group B receives a minimalistic voiding trial. In both groups the patient's catheter is removed at the operation room before returning to the gynecological ward.

Group A is the control group and presents the current procedures with strict voiding trial. Here, the patient will postoperatively try to void approximately every second hour after catheter removal or if she has sensation of bladder filling. The bladder is scanned before voiding to determine the bladder volume, and the voiding volume is measured. If the voiding volume is >150 ml and the residual volume is <200 ml, the patient can be discharged. If the patient cannot fulfill the criteria at the first voiding, the patient voids again 1 hour later and so on. If the residual volume is above 300 ml intermittent catheterization will be placed and the voiding trial regime restarts. If no acceptable residual volume is reached, the patient will be instructed in intermittent catheterization and there will be a postoperative follow-up the day after by telephone. If intermittent catheterization is not possible a closed catheter is placed which is opened approximately every third hour. The following day the patient will perform the voiding trial once again at the gynecological ward.

Group B is the intervention group with minimalistic voiding trial. The patients in this group need to have one spontaneous voiding before discharge with the sensation of normal voiding, meaning there is no measurement of the voiding volume or residual volume.

If the patients fail having spontaneous voiding or if the patients are in pain, the patients will undergo an ultrasound scanning to determine the bladder volume. If the patient's residual volume is above 400 ml the patient will be considered as failure and follow group A regime. If the patient's residual volume is under 400 ml the patient will continue group B regime and restart the regime.

To determine the development of postoperative urinary tract infection, urine retention and gynecological pain, the patients will have to answer a questionnaire when included in the study and two postoperative questionnaires at two weeks and three months after surgery. These questionnaires will be sent to e-box by using Open Redcap.

To assess the patients' need for guidance after surgery, the patients' calls to the gynecological ward after discharge will be registered.

Power calculation The sample size is calculated by means of medical-statistics.dk and the test 'comparing two-sample means'. Assuming the difference stated above, with a power of 80% we would need to allocate 84 patients (42 in each group) in the study. Estimating a drop-out rate of 10% we aim to include 47 in each group.

Inclusion criteria

* Patients who undergo anterior, posterior or vaginal vault prolapse surgery or bulking surgery at the departments of obstetric and gynecology, OUH.
* Patients who have the catheter removed at the operating room.
* Patients >18 years old.

Exclusion criteria

* Any surgery performed by due to malignancy
* Previous cancer in the pelvic area
* Previous radiation therapy in the pelvic area
* Previous surgery in the pelvic area
* Patients not understanding Danish
* Patients with mental or similar illness
* Patients with multiple sclerosis or diabetes type 1
* Patients with late KAD removal based on per operative assessment

Statistical analysis Descriptive statistics In the study the baseline data and characteristics will be reported as means or numbers with 95% confidence intervals with a significance level set at an alpha of 0,05. Differences between groups will be evaluated by Chi square or Fisher's exact test. When appropriate, unadjusted odds ratio's with 95% confidence intervals will be calculated.

Ethical consideration The study will be approved by Fortegnelse for Forskningsprojekter, Region of Southern Denmark.

The study will be conducted according to the principles of the Declaration of Helsinki II.

ELIGIBILITY:
Inclusion Criteria:

* • Women who undergo anterior, posterior or vaginal vault prolapse surgery or bulking surgery at the departments of obstetric and gynecology, OUH.

  * Women who have the catheter removed at the operating room.
  * Women >18 years old.

Exclusion Criteria:

* Any surgery performed by due to malignancy

  * Previous cancer in the pelvic area
  * Previous radiation therapy in the pelvic area
  * Previous surgery in the pelvic area
  * Patients not understanding Danish
  * Patients with mental or similar illness
  * Patients with multiple sclerosis or diabetes type 1
  * Patients with late KAD removal based on per operative assessment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Residual urine | 12 hours postoperatively
  Residual urine after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Martin Rudnicki, Principal Investigator — Odense Universitetshospital
Locations (1):
- martin Rudnicki, Odense C, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No
no plan